CLINICAL TRIAL: NCT04018703
Title: Effective Dose of Dexmedetomidine or Midazolam in Monitored Anesthesia Care for Patients Undergoing Ophthalmologic Surgery With Retrobulbar Nerve Block
Brief Title: The Study of Different Sedative Medications in Monitored Anesthesia Care During Eye Surgery With Local Anesthesia
Acronym: MAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Hui Qiao, Attending Anesthesiologist, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAC in Eye Surgery
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Balanced Anesthesia; Adjuvants,Anesthesia
Keywords: Monitored anesthesia care; Ophthalmic surgery; Dexmedetomidine; Midazolam
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine will be used for perioperative sedation.
  Interventions: Drug: Dexmedetomidine
- Midazolam (Experimental): Midazolam will be used for perioperative sedation.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — loading dose 0.5-2.5ug/kg followed by continuous infusion 0.2-0.5ug/kg/h
  Arms: Dexmedetomidine
Drug: Midazolam — loading dose 30-50ug/kg followed by continuous infusion 10-30ug/kg/h
  Arms: Midazolam

SUMMARY:
Due to the delicacy and long duration of the procedure, ophthalmic surgery put forward higher requirements to anesthesia management:

1. The patient with local anesthesia without sedation is in a state of awareness, which will cause intense stress resulting in increased blood pressure, heart rate, muscle tension and even sense of pain;
2. Traction of extraocular muscles and eyeballs can induce oculocardiac reflex, followed by bradycardia, atrial or ventricular arrhythmia, conduction block, and even more worsen, life-threatening cardiac arrest may occur;
3. With the increase in average life expectancy and the improvement of quality of life requirements, the number of elderly patients in ophthalmic surgery is also increasing. These elderly patients are often combined with hypertension, diabetes, etc. and decreased tolerance of with general anesthesia;
4. For some retinal detachment surgery with difficulty in resetting, the patients will be required to change to the prone position immediately after surgery to improve the success rate of resetting. Conventional general anesthesia management are cumbersome and costly, which may not be likely to achieve the swift emergence.

Nowadays, monitoring Anesthesia Care (MAC) has developed into a flexible and unique anesthesia technology combining intravenous anesthesia with regional block anesthesia. MAC provides reasonable balance between economy, comfort and safety, efficiency by continuous monitoring of changes in respiratory and circulatory system, during process of sedation and analgesia. Airway management will be another issue as surgeons operate on the side of head and face. Studies have shown that MAC can achieve adequate sedation and analgesia to decrease blood pressure, provide acceptable surgical fields and reduce adverse reactions such as perioperative stress, pain and anxiety. Meanwhile, MAC make patients comfortable enough to cooperate with the surgeons, easy to be awakened with relatively short operation duration and improvement of perioperative safety.

DETAILED DESCRIPTION:
The allocation sequence is generated by computer random number generation, and the allocation is placed in sequentially numbered opaque sealed envelopes by a non-investigator. Enrolment and data collection are performed by trained research staff who are not involved in the care of the patients. The treating clinicians are not possible to be blinded to the assignment group, but all other staff involved in both the collection and collation of data, and administration of neurocognitive testing, are blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for ophthalmic surgery with retrobulbar nerve block

Exclusion Criteria:

* Patients with severe cardiac, pulmonary, hepatic, or renal dysfunction. Patients with a preoperative history of mental disorder, hearing disorder, II-III degree atrioventricular block, known allergy or hypersensitivity to a2 receptor agonists and refusal of (or contraindications to) PNB. Patients with anticipated difficult airway.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative change of Observer's Assessment of Alertness/Sedation scale (OAA/S) | OAA/S score will be recorded from patient arrival in the operating room to about 30 minutes after surgery at following time points: before sedative administration, before skin incision, every 5 minutes intraoperatively and every 10 minutes in PACU.
  Conventional subjective sedation scales with 1 to 5. Successful sedation was defined as an OAA/S scale score between 1 and 3, while failure was defined as an OAA/S score of more than 3.
Numerical rating scale (NRS) | Immediately after surgery, the surgeons report NRS only once
  The surgeons rated anesthesia management on a numerical rating scale (NRS), ranging from 0 to 10, with 10 defined as the best condition and 0 as the worst.

SECONDARY OUTCOMES:
Intraocular pressure | Intraocular pressure will be measured at two time points: before sedative medication administration and before skin incision.
  Measured with Tono-Pen tonometer
Bispectral index (BIS) | Bis will be continuously recorded with BIS monitor from arrival in the operating room to discharge to ward (about 30 minutes after surgery).
  Anesthesia depth index
Visual analogue scale (VAS) | VAS will be recorded at the following time points until 1h postoperatively: before sedative medication administration, before skin incision, every 10 minutes intraoperatively and 1h postoperatively
  Patient self-report pain score ranging from 0 to 10, with 0 defined as no pain at all and 10 as the intolerable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Wenxian Li, M.D. Ph.D., Study Director — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye, Ear, Nose and Throat Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No